CLINICAL TRIAL: NCT01877733
Title: Effective Rehabilitation of Patients Operated With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/1678
Record Dates: First submitted 2013-04-16; First posted 2013-06-14 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis
Keywords: Resistance training
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximal strenght training (Experimental): Training maximal strength training 3 times a week/1 physiotherapy session for 8 weeks
  Interventions: Other: Maximal strength training
- Standard rehabilitation (No Intervention): 2-3 physiotherapy sessions a week for 8 weeks/telephone contact by project leader once a week/writing training diary

INTERVENTIONS:
Other: Maximal strength training
  Arms: Maximal strenght training

SUMMARY:
The purpose of this study is to investigate the effect of maximal strength training (MST) compared to standard rehabilitation in patients operated with total knee arthroplasty. Previous studies report reduced physical function and muscle strength despite successful surgery inserting an artificial implant.

Furthermore, great loss of muscle strength has been found in these patients in the early postoperative phase.

The study is a randomized controlled trial. The investigators hypothesize that MST will increase muscle strength and physical function more than standard rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* unilateral osteoarthritis,
* < 75 years

Exclusion Criteria:

* disease(s) that compromise testing/training,
* unable to understand written and verbal instructions and information,
* osteoarthritis in the contralateral leg that needs treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Muscle strength in leg extension and leg press | Measured preoperatively, after 7 days, 10 wks and 1 year
  Measured preoperatively implies measuring the outcome within the last month prior to surgery

SECONDARY OUTCOMES:
6 minute walk test | preopertively, 7 days postoperatively and after 1 year
  Measuring the outcome preoperatively implies testing within the last month prior to surgery
KOOS; Knee injury and osteosarthritis outcome score | Preoperatively (within 1 month prior to surgery), 7 days postoperatively and 10 wks and 1 year postoperatively
EQ-5D (measure of health outcome) | Preoperatively (within 1 month prior to surgery), 7 days, 10 wks and 1 year postoperatively
VAS scale recording pain | preoperatively (within 1 month prior to surgery), 7 days, 10 wks and 1 year postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vigdis S Husby, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Husby VS, Foss OA, Husby OS, Winther SB. Randomized controlled trial of maximal strength training vs. standard rehabilitation following total knee arthroplasty. Eur J Phys Rehabil Med. 2018 Jun;54(3):371-379. doi: 10.23736/S1973-9087.17.04712-8. Epub 2017 Sep 13. PMID 28901118
- [Result] Winther SB, Foss OA, Klaksvik J, Husby VS. Pain and load progression following an early maximal strength training program in total hip- and knee arthroplasty patients. J Orthop Surg (Hong Kong). 2020 Jan-Apr;28(2):2309499020916392. doi: 10.1177/2309499020916392. PMID 32301372